CLINICAL TRIAL: NCT04397796
Title: Phase 1b Randomized, Double-Blind, Placebo-Controlled Study Of The Safety Of Therapeutic Treatment With Immunomodulatory Mesenchymal Stem Cells In Adults With COVID-19 Infection Requiring Mechanical Ventilation
Brief Title: Study of the Safety of Therapeutic Tx With Immunomodulatory MSC in Adults With COVID-19 Infection Requiring Mechanical Ventilation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QUILT-COVID-19-MSC
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-04

CONDITIONS: COVID
Keywords: IMMUNOMODULATORY MESENCHYMAL STEM CELLS; MSC; COVID-19; Mechanical ventilation; Severe respiratory distress
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BM-Allo.MSC (Experimental): Subjects in the experimental arm will be administered BM-Allo.MSC
  Interventions: Biological: BM-Allo.MSC
- Placebo (Placebo Comparator): Subjects in the control arm will be treated with placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BM-Allo.MSC — BM-Allo.MSC for Infusion, is manufactured from normal donor derived bone marrow product and are phenotypically CD73+, CD90+, CD105+, and negative for CD14-, CD34-, CD45-, HLA-DR-.
  Arms: BM-Allo.MSC
Biological: Placebo — plasmalyte and human albumin
  Arms: Placebo

SUMMARY:
This is a phase 1b randomized, double-blind, placebo-controlled study in adult subjects with Coronavirus Disease 2019 (COVID-19). This clinical trial will evaluate the preliminary safety and efficacy of BM-Allo.MSC vs placebo in treating subjects with severe disease requiring ventilator support during COVID 19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines. For subjects that are intubated and/or sedated, or otherwise unable to provide consent, prospective consent from a legally-authorized representative is required. The subject or his/her legally authorized representative must be able to provide consent.
3. Has laboratory-confirmed positive novel coronavirus (SARS-CoV-2) test, as determined by polymerase chain reaction (PCR), or other commercial or public health assay in any specimen < 72 hours prior to enrollment, or meets the criteria to guide the evaluation and testing of patients under investigation (PUI) for COVID-19 (https://emergency.cdc.gov/han/2020/HAN00428.asp).
4. Requiring mechanical ventilatory support with moderate to severe Acute Respiratory Distress Syndrome (ARDS) as determined by the Berlin criteria:

   1. Bilateral opacities present on a chest radiograph or computed tomographic (CT) scan. These opacities are not fully explained by pleural effusions, lobar collapse, lung collapse, or pulmonary nodules.
   2. Origin of Edema: Respiratory failure not fully explained by cardiac failure or fluid overload.
   3. Oxygenation: Moderate to severe impairment of oxygenation must be present, as defined by the ratio of arterial oxygen tension to fraction of inspired oxygen (PaO2/FiO2). The severity of the hypoxemia defines the severity of the ARDS:

      * Moderate: PaO2/FiO2 >100 mmHg and ≤ 200 mmHg, on ventilator settings that include PEEP ≥ 5 cm H2O
      * Severe: PaO2/FiO2 ≤100 mmHg on ventilator settings that include PEEP ≥5 cm H2O Subjects receiving extracorporeal membrane oxygenation (ECMO) will not be enrolled in this study.
5. High-sensitivity C-reactive Protein (hs-CRP) serum level > 4.0 mg/dL
6. Acute Physiology and Chronic Health Evaluation (APACHE IV) score > 5
7. Agrees to the collection of nasopharyngeal (NP) swabs and venous blood per protocol.
8. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
9. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception while on study and for at least 1 month after the last dose of BM-Allo.MSC. Non-sterile male subjects must agree to use a condom while on study and for up to 1 month after the dose of BM-Allo.MSC. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), oral contraceptives, and abstinence.

Exclusion Criteria:

1. Known hypersensitivity to any component of the study medication(s).
2. Signs of multisystem organ failure. Liver function tests (LFTs) > 5x normal.
3. Intubated > 72 continuous hours.
4. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
5. Pregnant and nursing women. A negative serum pregnancy test during screening (within 72 hours prior to the first dose) must be documented before MSCs are administered to a female subject of child-bearing potential.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Francis Medical Center, Lynwood, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BM-Allo.MSC: Subjects in the experimental arm will be administered BM-Allo.MSC
  BM-Allo.MSC: BM-Allo.MSC for Infusion is manufactured from normal donor derived bone marrow product and are phenotypically CD73+, CD90+, CD105+, and negative for CD14-, CD34-, CD45-, HLA-DR-.
Period: Overall Study
Arm/Group | BM-Allo.MSC | Placebo
Started | 3 | 1
Completed | 0 | 0
Not Completed | 3 | 1
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BM-Allo.MSC | Placebo | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.5) | 64.0 | 62.8 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Subjects with severe disease requiring ventilator support during COVID-19 infection [Count of Participants; unit: Participants] | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Within 30 Days of Randomization
Description: Incidence of AEs within 30 days of randomization.
Time Frame: 30 days
Population: Analysis population is all randomized subjects who received at least one dose of study intervention (safety analysis population)
Measure: Count of Participants; unit: Participants
Arm/Group | BM-Allo.MSC | Placebo
Number analyzed (Participants) | 3 | 1
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: From randomization through 30 days past the last dose, up to 34 days.
Arm/Group | BM-Allo.MSC | Placebo
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BM-Allo.MSC (N=3) | Placebo (N=1)
Disease progression (General disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BM-Allo.MSC (N=3) | Placebo (N=1)
Disease progression (General disorders) | 3 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Ear injury (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Obstructive shock (Vascular disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Endotracheal intubation (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
The study is terminated early due to low enrollment. Efficacy of the Investigational Product is not analyzed.

Race was not collected in the CRFs for subjects and therefore is not presented in the data output for these subjects.

Treatment-Emergent Adverse Events Table includes Serious Adverse Events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT04397796/Prot_SAP_000.pdf